CLINICAL TRIAL: NCT01152593
Title: Effect of Intranasal Mupirocin on Rate of Staphylococcus Aureus Surgical Site Infection Following Cesarean Sections
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Gai Shrem, MD, Hillel Yaffe Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HYMC0033-10
Record Dates: First submitted 2010-05-31; First posted 2010-06-29 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2010-06

CONDITIONS: Surgical Wound Infection; Cesarean Section; Staphylococcus Aureus
MeSH Terms: conditions — Surgical Wound Infection; Staphylococcal Infections | interventions — Mupirocin

ARMS (1):
- Intranasal Mupirocin (Experimental)
  Interventions: Drug: Mupirocin

INTERVENTIONS:
Drug: Mupirocin — Intranasal cream given to patient after confirmation of colonization

SUMMARY:
The investigators believe that irradication of nose colonization of staphyloccocus aureus will reduce the incidence of surgical site infections after cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Women assigned to undergo cesarean section

Exclusion Criteria:

* All others

Sex: Female
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2010-07; Primary Completion 2014-07 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Reduction of the incidence of surgical site infections after cesarean section | Four years

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel